CLINICAL TRIAL: NCT04708340
Title: A Two-part, Two-cohort, Double-blind, Randomized, Placebo-controlled, Multicenter Phase 1/2 Study to Evaluate the Safety, Tolerability and Efficacy of REJUVEINIX (RJX) in Patients With COVID-19
Brief Title: Tolerability and Efficacy of RJX in Patients With COVID-19
Acronym: RJX
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RPI015
Record Dates: First submitted 2021-01-04; First posted 2021-01-13 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: COVID-19; Acute Respiratory Distress Syndrome; SARS-CoV-2; Hypoxemia
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome; Hypoxia | interventions — ascorbic acid, magnesium sulfate heptahydrate, cyanocobalamin, thiamine hydrochloride, riboflavin 5' phosphate, niacinamide, pyridoxine hydrochloride, and calcium D-pantothenate drug combination; Sodium Chloride; Water; Injections; Saline Solution

STUDY DESIGN:
Intervention Model Description: In Part 1, RJX will be administered daily for 7 days (1 cycle). In Part 2, Placebo or RJX will be administered daily for 7 days for 1 cycle but may receive 2 cycles.
  Each Cohort is comprised of Part 1, a single site, and Part 2, multiple sites. The 2 Cohorts are:
  Cohort 1:
  * Hospitalized COVID-19 patients ≥18 years without hypoxemia and either not receiving any oxygen therapy OR are receiving supplemental oxygen via mask or nasal prongs (clinical status score 4 or 5 on 8-point ordinal scale).
  * Patients are required to have the following high-risk characteristics
    * Age ≥65 years AND type 2 diabetes or hypertension OR
    * Age ≥18 years with abnormal blood tests AND CRP >50 mg/L PLUS at least 1 of the following biomarkers abnormal: a. D-dimer, b. Ferritin, c. High sensitivity cardiac troponin, d. LDH
  Cohort 2:
  • Hospitalized COVID-19 patients with hypoxemia and without ARDS who are receiving either non-invasive positive pressure ventilation (NIPPV) OR high flow oxygen
Who Masked: Participant, Investigator
Masking Description: Masking the dose administered
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: RJX (Active Comparator): 1. RJX 20 mL (10 mL of Vial A plus 10 mL of Vial B) mixed in normal saline, total volume 120 mL, administered by IV infusion over a period of 40 minutes +/- 10 minutes once daily.
  2. Standard of care (current antiviral and/or supportive care treatment currently in place at the institution for COVID-19 treatment).
  3. Patients in Part 1 are allowed to receive only one 7-day cycle of RJX while patients in Part 2 may be treated daily for up to 14 days.
  Interventions: Drug: Rejuveinix (RJX) Active Comparator
- Arm B: Placebo (Placebo Comparator): 1. Placebo (total of 20 mL normal saline) mixed in normal saline IV, total volume 120 mL of normal saline IV, administered by IV infusion over a period of 40 minutes +/- 10 minutes once daily.
  2. Standard of care (current antiviral and/or supportive care treatment currently in place at the institution for COVID-19 treatment).
  3. Patients in Part 1 will not receive placebo.
  4. Patients in Part 2 may be treated daily for up to 14 days.
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Rejuveinix (RJX) Active Comparator — Active drug comprised of: ascorbic acid, magnesium sulfate heptahydrate, cyanocobalamin, thiamine, riboflavin 5' phosphate, niacinamide, pyridoxine, calcium d-pantothenate, and sodium bicarbonate.
  Other Names: RJX; Rejuveinix
  Arms: Arm A: RJX
Drug: Placebo Comparator — 0.9% Sodium Chloride in Water for Injection a.k.a. Normal Saline for injection
  Other Names: 0.9% Sodium Chloride in Water for Injection, USP.; Normal Saline for Injection, USP
  Arms: Arm B: Placebo

SUMMARY:
This study is designed as a 2-part, 2-cohort, double-blind, randomized, placebo controlled, multicenter Phase 1/2 study to evaluate the safety, tolerability and efficacy of RJX in patients with COVID-19.

DETAILED DESCRIPTION:
For each cohort, there will be an open label Safety Lead-in (Part 1) and a placebo controlled, randomized, double-blind portion (Part 2). In Part 1, RJX will be administered daily for 7 days. In the active treatment arm of Part 2 for both cohorts, RJX will be administered daily for 7 days per cycle and patients may receive up to 2 cycles. As detailed below, patients will be allowed to receive a second 7 day cycle of therapy based on the medical judgment of the Investigator. The total RJX exposure during Part 2 could therefore be up to 14 days. Both cohorts will start and enroll in parallel and independently. A safety follow-up period will begin at Day 14/Discharge, or when treatment is discontinued, and will continue for approximately 60 days post discharge. Part 1 will be conducted at a single site and Part 2 will be conducted at multiple sites. The 2 cohorts in this study are:

* Cohort 1:

  * Hospitalized COVID-19 patients ≥18 years without hypoxemia who are either not receiving any oxygen therapy OR are receiving supplemental oxygen via mask or nasal prongs (namely, clinical status score 4 or 5 on an 8-point ordinal scale).
  * Patients are required to have the following high-risk characteristics

    1. Age ≥65 years AND type 2 diabetes or hypertension OR
    2. Age ≥18 years with abnormal blood tests AND CRP >50 mg/L PLUS at least 1 of the following biomarkers:

       1. D-dimer >1,000 ng/mL,
       2. Ferritin >500 µg/L,
       3. High sensitivity cardiac troponin >2 × upper limit of normal (ULN),
       4. LDH >245 U/L.
* Cohort 2:

  * Hospitalized COVID-19 patients with hypoxemia without ARDS who are receiving either non-invasive positive pressure ventilation (NIPPV) OR high flow oxygen (namely, clinical status score 3 on an 8-point ordinal scale).

ELIGIBILITY:
Inclusion Criteria

Cohort 1 (Part 1 and Part 2):

1. Hospitalized COVID-19 patients ≥18 years without hypoxemia who are either not receiving any oxygen therapy OR are receiving supplemental oxygen via mask or nasal prongs (namely, clinical status score 4 or 5 on an 8-point ordinal scale)
2. Hospitalized COVID-19 patients age ≥65 years AND type 2 diabetes or hypertension, OR
3. Hospitalized COVID-19 patients ≥18 years AND abnormal blood tests with CRP >50 mg/L PLUS at least 1 of the following biomarkers:

   1. D-dimer >1,000 ng/mL
   2. Ferritin >500 µg/L
   3. High sensitivity cardiac troponin >2 × ULN
   4. LDH >245 U/L

   Cohort 2 (Part 1 and Part 2):
4. Hospitalized COVID-19 patients with hypoxemia who are either receiving NIPPV OR high-flow oxygen (namely, clinical status score 3 on an 8-point ordinal scale).
5. Bilateral opacities on a chest x-ray OR chest CT scan. Cohort 1 and Cohort 2 (Parts 1 and 2)
6. Male and non-pregnant, non-lactating female patients with SARS-CoV-2 infection that is documented by a Food and Drug Administration (FDA)-authorized diagnostic reverse transcription polymerase chain reaction test at/or within 4 days of Screening
7. ≥18 years of age
8. Body weight ≥40 kg at Screening
9. History of COVID-19 within the last 2 weeks prior to study enrollment
10. The patient OR a legally authorized representative has provided written informed consent
11. Females of childbearing potential must have a negative beta human chorionic gonadotropin pregnancy test at Screening
12. Females of childbearing potential must agree to be abstinent or else use a medically acceptable form of contraception from the Screening period through Day 28. Medically acceptable forms of contraception including implants, injectables, combined oral contraceptives, some intrauterine devices, sexual abstinence or vasectomy, and double-barrier method [condom and occlusive cap (diaphragm or cervical/vault caps)] with spermicidal foam/gel/film/suppository

Exclusion Criteria Cohort 1

1. Receiving high-flow oxygen OR NIPPV. Cohort 1 and Cohort 2
2. ARDS by Berlin definition (Appendix 16.2)
3. On extracorporeal membrane oxygenation
4. Uncontrolled hypertension (systolic blood pressure [BP] >150 mmHg and/or diastolic BP >100 mmHg), unstable angina, congestive heart failure of New York Heart Association Classification Class III or IV (i.e., Class III: marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g., walking short distances [20 100 m], comfortable only at rest; Class IV: severe limitations, experiences symptoms even while at rest, mostly bedbound patients), serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infarction within 12 months prior to enrollment
5. Subjects with a history of congenital long QT syndrome or of Torsades de pointes; subjects with bradycardia (<60 bpm), heart block (excluding 1st degree block, being PR interval prolongation only); subjects with any of the following findings on electrocardiogram (ECG): QTc interval >470 msec in women OR >450 msec in men; subjects requiring any drugs known to prolong the QTc interval, including antiarrhythmic medications
6. Shock or hypotension requiring vasoactive peptides, such as dopamine, norepinephrine, epinephrine, or dobutamine
7. Renal function impairment with creatinine ≥2 mg/dL
8. Liver function impairment with total bilirubin ≥2 mg/dL
9. Platelet count <50,000/µL
10. Multi-organ failure
11. History of an allergic reaction or hypersensitivity to the study drug or any component of the study drug formulation
12. Use of systemic corticosteroids, nonsteroidal anti-inflammatory drugs, antibiotics, and antiviral drugs that are not part of the standard of care
13. Presence of any uncontrolled concomitant illness (e.g., bacterial sepsis or invasive fungal infection), or other serious illness and medical conditions, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with their participation in the study
14. Pregnancy or breast-feeding (for women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Safety as measured by DLTs and drug related SAE's | Up to 60 days post-enrollment
  • Part 1, Cohorts 1 and 2: Cumulative incidence of DLTs and drug-related SAEs (viz., sum of DLT + SAEs) reported within 14 days of first dose of RJX (Part 1) or reported within 60 days of first dose of study drug (Part 2)
Tolerability and Efficacy measured by progression of disease through an ordinal scale. | Within 2 weeks
  • Part 2, Cohort 1: Progression to severe disease on an 8-point ordinal scale from a clinical status score of 4 or 5 to a clinical status score of 3, 2, or 1 within 2 weeks of first dose of study drug
Efficacy measured by time to resolution of respiratory failure | 60-days post enrollment
  • Part 2, Cohort 2: Time to resolution of respiratory failure (TTRRF), with status change on an 8-point ordinal scale from a clinical status score of 3 to a clinical status score of ≥4

SECONDARY OUTCOMES:
Efficacy as measured by day of ICU care. | 60-days post enrollment
  The key secondary endpoints for Parts 1 and 2, Cohorts 1 and 2 are:
  • Mean number of days of ICU care
Safety, Tolerability, Efficacy measured by mortality over 28 Days. | 28-days post enrollment
  The key secondary endpoints for Parts 1 and 2, Cohorts 1 and 2 are:
  • Proportion of patients that die (any cause) by Day 28 post randomization (patient may be inpatient or outpatient in follow up)
Efficacy measured by mean change in baseline clinical status on Days 7 and 14. | 14-days post enrollment
  Additional secondary endpoint for Parts 1 and 2, Cohorts 1 and 2 are:
  • Mean change from baseline of clinical status using an 8-point ordinal scale (with 8 being "Not hospitalized, no limitations on activities", and 1 being "Death") at Days 7 and 14
Efficacy measured by mean change in hospitalization days on Days 7 and 14. | 14-days post enrollment
  Additional secondary endpoint for Parts 1 and 2, Cohorts 1 and 2 are:
  • Mean number of hospitalization days
Efficacy measured by time to coming off supplemental oxygen on Days 7 and 14. | 14-days post enrollment
  Additional secondary endpoint for Parts 1 and 2, Cohorts 1 and 2 are:
  • Time to coming off supplemental oxygen (defined as a score of ≥5 on an 8-point ordinal scale; Cohort 1 only)
Safety and Efficacy measured by time from first dose to renal therapy. | 60-days post enrollment
  Additional secondary endpoint for Cohort 2, Part 2 is:
  • Time to initiation of renal replacement therapy

OTHER OUTCOMES:
Evaluate Change in Serum CRP Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of CRP (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum Ferritin Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of ferritin (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum D-dimer Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of D-dimer (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum LDH Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of LDH (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum IL-6 Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of IL-6 (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum IL-10 Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of IL-10 (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum TNF-α Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of TNF-α (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum TGF-β Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of TGF-β (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum C3 Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of C3 (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Serum C5 Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of C5 (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in Plasma ascorbic acid Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of ascorbic acid (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in plasma niacinamide Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of niacinamide (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in plasma thiamine Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of thiamine (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.
Evaluate Change in plasma cyanocobalamin Concentration | Up to 28-days post randomization
  The exploratory endpoint for Parts 1 and 2 is:
  Kinetic of response of cyanocobalamin (comparison of baseline to Day 7, Day 14, and Day 28 post-randomization). These laboratory measures will be obtained either as an inpatient or an outpatient follow-up.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - Memorial Hermann Southeast Hospital, Houston, Texas
  - Christus Santa Rosa Hospital, New Braunfels, Texas

IPD SHARING:
Plan to Share IPD: No